CLINICAL TRIAL: NCT01618383
Title: Study of the Enteric Nervous System Using Colonic Biopsies in Parkinson Patients With LRRK2 Mutation
Acronym: EnteroLarc
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of patients
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC11_0110
Record Dates: First submitted 2012-06-11; First posted 2012-06-13 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; gut; colon; biopsies; LRRK2
MeSH Terms: conditions — Parkinson Disease | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Colonic biopsies (Other): Colonic biopsies obtained during the course of colonoscopy or rectosigmoidoscopy
  Interventions: Other: colonoscopy or rectosigmoidoscopy

INTERVENTIONS:
Other: colonoscopy or rectosigmoidoscopy — Usual procedure

SUMMARY:
The clinical and pathological similarities between LRRK2 related parkinsonism and idiopathic Parkinson's disease (PD) indicate that monogenetic LRRK2 parkinsonism may be a paradigm for the development of Lewy bodies disease, and a careful look at discrepancies between these two conditions may provide insight into the pathogenesis of PD. The early involvement of the enteric nervous system (ENS) during PD led to theories that an as yet unidentified external agent entering the ENS causes PD . If lesions of the ENS are found in patients who present with a genetic form of parkinsonism would go against this notion, and thus provide insight to the pathophysiology of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 30-80, both genders
* Parkinson's disease patients
* Parkinson's disease patients with G2019S mutations
* Controls: patient at risk of colic cancer for whom a coloscopy is required

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Presence of alpha-synuclein aggregates in colonic biopsies using immunohistochemistry | 3 months

SECONDARY OUTCOMES:
Analysis of intestinal permeability in biopsies using Ussing's chambers | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Tiphaine ROUAUD, Doctor, Principal Investigator — Nantes University Hospital
Locations (1):
- University Hospital, Nantes, France